CLINICAL TRIAL: NCT02296606
Title: Interrater Reliability of Subjective Pupillary Assessments
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, DaiWai Olson, Associate Faculty, University of Texas Southwestern Medical Center
Other Study IDs: STU042014-043
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Interrater Reliability Among Pupillary Assessments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, observational, non-randomized study of interrater reliability of pupillary assessments, comparing two clinical assessments to the Pupillometer.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for this study if they have been diagnosed with some form of brain trauma (e.g., stroke, traumatic brain injury, aneurysm)

Exclusion Criteria:

* Prisoners
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for the study are those that have been diagnosed some form of brain trauma where brain swelling has been identified and pupil dilation has been incorporated into standard of care (e.g., TBI, stroke).
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants underwent three pupil exams, two by flashlight/pen light by two different assessors, and one by a researcher using the Pupillometer Device. Pupil exams occurred up to three times daily for the extent that the patient was in the ICU at the enrolling hospital.
Period: Overall Study
Arm/Group | All Participants
Started | 127
Completed | 127
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 103
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 127

OUTCOME MEASURES:

1. Primary Outcome: 1. Explore the Interrater Reliability of Pupillary Assessments When Conducted in the Natural Setting by a Diverse Group of Practitioners
Description: Two human assessors conducted and recorded the results of a clinical pupillary assessment on one patient within 5 minutes of one another. The researcher then conducted and recorded pupillary information on the same patient (within the same 5 minute window) using the NeurOptics Pupillometer.
Time Frame: 9 months of pupillary assessments
Measure: Mean (95% Confidence Interval); unit: Kappa score
Units Other Than Participants: paired pupil assessments
Groups:
- All Participants: There are no groups/arms for the purpose of this study.
Arm/Group | All Participants
Number analyzed (Participants) | 127
Number analyzed (paired pupil assessments) | 2329
Kappa score | .54 [.50 to .57]

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No